CLINICAL TRIAL: NCT03555695
Title: Karate Intervention to Change Kinematic Outcomes in Parkinson's Disease
Brief Title: Kick Out Parkinson's Disease- Karate Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18012313
Record Dates: First submitted 2018-05-30; First posted 2018-06-13 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease
Keywords: karate; exercise
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a non-randomized, open-label, non-blinded, 10-week pilot study of a novel intervention, namely, non-contact karate, for early to middle stage PD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Karate Class Participants (Experimental): Eligible subjects will engage in twice-weekly karate classes for 10 weeks, specifically designed for individuals with early to middle stage PD. Subjects will also complete an in-person pre-intervention focus group and post-intervention focus group, as well as a 6 month post-intervention follow up phone call.
  Interventions: Behavioral: Karate Classes; Behavioral: Pre-Intervention Focus Group; Behavioral: Post-Intervention Focus Group

INTERVENTIONS:
Behavioral: Karate Classes — Eligible subjects will engage in twice-weekly karate classes for 10 weeks, specifically designed for individuals with early to middle stage PD, focused on incorporating upper and lower limb movements in multiple directions, increasing awareness throughout the body, shifting body weight and rotation, relaxation of the muscles, improving reaction time, using complex repetitive actions to improve coordination, footwork training and centered weight shifts to help with fall prevention, and striking shields for self-defense and stress relief.
Behavioral: Pre-Intervention Focus Group — At the pre-intervention focus group, the study logistics will be reviewed, informed consent process will occur, the subject will complete a brief, individual pre-intervention assessment focused on overall mobility, gait, balance, mood, neurological status, and quality of life, and the subjects will be prompted to share aloud their thoughts on exercise, balance, and mindfulness practices in general and in PD specifically, and any expectations or preconceptions that they have regarding karate classes for PD.
Behavioral: Post-Intervention Focus Group — At the post-intervention focus group, the pre-intervention assessments will be readministered, along with an assessment of the subject's global impression of change. Subjects will be prompted to share their thoughts on how the intervention impacted their overall wellbeing, balance, and mindfulness; whether the intervention achieved their expectations; and they will be asked to provide feedback for improvements.

SUMMARY:
The benefits of exercise for general health and wellbeing in older adults are well-established. Balance exercises such as tai chi and yoga, along with resistance training, can improve or maintain physical function in older adults and enhance muscle strength. Furthermore, aerobic activity is critical for maintaining and improving cardiovascular and functional health. Noncontact boxing has recently seen a surge in popularity among individuals with Parkinson's Disease (PD), with components of both aerobic and balance exercise. While participants anecdotally note improvements in stress and physical function, this has only been minimally studied. However, drawing on this experience and the combined aerobic, balance, and mindfulness practices that comprise karate, we hypothesize that participation in structured karate programs may offer similar or greater benefits. Specifically, the aim of this study is to test whether and to what degree a community-based karate class tailored for individuals with early- to middle-stage Parkinson's Disease (PD) 1) is feasible; and 2) improves objective and patient-reported outcomes.

DETAILED DESCRIPTION:
For 10 weeks, eligible subjects will engage in twice-weekly karate classes, specifically designed for individuals with early to middle stage PD, focused on incorporating upper and lower limb movements in multiple directions, increasing awareness throughout the body, shifting body weight and rotation, relaxation of the muscles, improving reaction time, using complex repetitive actions to improve coordination, footwork training and centered weight shifts to help with fall prevention, and striking shields for self-defense and stress relief.

Before beginning the karate classes, each subject will attend a pre-intervention focus group during which subjects will complete an assessment focused on overall mobility, gait, balance, mood, and quality of life. Subjects will be prompted to share their thoughts on exercise, balance, and mindfulness practices in general and in PD specifically.

Following the 10 weeks of twice-weekly karate classes, subjects will attend a post-intervention assessment and focus group during which the pre-intervention assessments will be repeated and the subject's impressions about the karate classes and their effectiveness will be measured.

Finally, the study team will contact subjects 6 months post-intervention to assess continued engagement in karate or related activities and again, the subject's quality of life and global impression of change.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be those diagnosed with Parkinson's Disease by a treating neurologist; if the subject is seen at Rush University Medical Center, this will be verified via chart review. If the subject is seen elsewhere, he or she will be asked to have their neurologist sign a form confirming the diagnosis of Parkinson's Disease and indicating the subject's HY stage (with definitions of each stage provided on the form for providers who may not be familiar with HY staging) at the most recent visit, to be sent back to the study coordinator for eligibility verification.
* English speaking
* Living within the Chicago area
* Subjects may be untreated for Parkinson's Disease, or may be taking any individual PD medication or combination thereof. Subjects may or may not have had Deep Brain Stimulation. Subjects may or may not be receiving physical or occupational therapy. Subjects will be encouraged to maintain their same medication regimen throughout the duration of the 10-week study, however if emergent issues arise requiring medication changes, the subject will not be disqualified.

Exclusion Criteria:

* Subjects requiring an assistive device (cane, walker, wheelchair) or the assistance of another person in order to ambulate.
* Subjects with active psychosis or exhibiting symptoms of a severe psychiatric disorder.
* Subjects unable to commit to attending, or to travel to, two classes weekly for 10 weeks.
* Subjects previously participating in a karate or other martial arts program, including boxing programs for PD, in the past 30 days.
* Subjects with atypical parkinsonism, including Progressive Supranuclear Palsy, Multiple System Atrophy, Dementia with Lewy Bodies, Corticobasal Syndrome, drug-induced parkinsonism, vascular parkinsonism, or atypical parkinsonism not otherwise specified, according to the referring neurologist.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jori Fleisher, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Fleisher JE, Sennott BJ, Myrick E, Niemet CJ, Lee M, Whitelock CM, Sanghvi M, Liu Y, Ouyang B, Hall DA, Comella CL, Chodosh J. KICK OUT PD: Feasibility and quality of life in the pilot karate intervention to change kinematic outcomes in Parkinson's Disease. PLoS One. 2020 Sep 9;15(9):e0237777. doi: 10.1371/journal.pone.0237777. eCollection 2020. PMID 32903267

RESULTS

PARTICIPANT FLOW:
Groups:
- Karate Class Participants: Eligible subjects will engage in twice-weekly karate classes for 10 weeks, specifically designed for individuals with early to middle stage PD. Subjects will complete in-person pre- and post-intervention focus groups, and a 6 month post-intervention follow up phone call.
  Pre-Intervention Focus Group: Study logistics will be reviewed, informed consent process will occur, the subject will complete a brief, individual pre-intervention assessment focused on overall mobility, gait, balance, mood, neurological status, and quality of life. Subjects will be prompted to share their thoughts on exercise, balance, and mindfulness practices in general and in PD specifically, and any expectations they have regarding karate for PD.
  Karate Classes: Specifically designed for individuals with early to middle stage PD, focused on incorporating limb movements in multiple directions, increasing body awareness, shifting body weight and rotation, muscle relaxation, improving reaction time, using complex repetitive actions to improve coordination, footwork training and centered weight shifts to help with fall prevention, and striking shields for self-defense and stress relief.
  Post-Intervention Focus Group: Pre-intervention assessments will be readministered, along with global impression of change. Subjects will be asked their thoughts on how the intervention impacted overall wellbeing, balance, and mindfulness; whether the intervention met their expectations; and to provide feedback.
Period: Overall Study
Arm/Group | Karate Class Participants
Started | 19
Completed | 15
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1
Not completed — appendicitis (unrelated) | 1
Not completed — pre-existing sciatica | 1

BASELINE CHARACTERISTICS:
Arm/Group | Karate Class Participants
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 19
Timed Up and Go [Mean (Standard Deviation); unit: Seconds] | 9.6 (2.23)
Parkinson's disease Quality of Life-short form [Mean (Standard Deviation); unit: units on a scale] — Validated eight-item measure, range 0-100, where lower scores indicate better quality of life
  units on a scale | 25.3 (20.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mobility as Measured by the Timed Up & Go (TUG)
Description: The Timed Up & Go (TUG) is a well-validated, brief measure of mobility. To complete this assessment, subjects sit in a standard arm chair and are instructed that when the team member says "Go", they should stand up from the chair, walk at their normal pace to a taped line, turn, walk back to their chair at a normal pace, and sit down again. The study team member will record the TUG results in seconds using a stopwatch. A lower TUG result indicates greater mobility. Scores at the pre- and post-intervention focus groups will be compared.
Time Frame: 10 weeks
Population: 15/19 participants completed the 10-week intervention
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Karate Class Participants
Number analyzed (Participants) | 15
seconds | 9.0 (1.89)
Statistical Analysis 1: Comparison: Karate Class Participants; Test type: Superiority; p = 0.12, t-test, 2 sided; Mean Difference (Final Values) = 0.6

2. Secondary Outcome: Change in Overall Well-being as Measured by the Patient Global Impression of Change Scale (PGIC)
Description: The Patient Global Impression of Change Scale (PGIC) is a single-item rating scale that asks subjects to rate their overall response to the intervention using a 7-point rating scale. Percentages of subjects endorsing each of the 7 response options will be compared. This scale will be completed at the post-intervention focus group.
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Karate Class Participants
Number analyzed (Participants) | 15
Participants
  "Almost the same" | 1
  "A little better" | 1
  "Moderately better" | 8
  "Better, definite improvement" | 4
  "Great deal better" | 1

3. Secondary Outcome: Quality of Life - Parkinson's Disease Questionnaire Short Form (PDQ-8)
Description: Validated 8-item PD-specific health-related quality of life measure; lower scores (score range 0-100) indicate better quality of life
Time Frame: 10 weeks
Population: 15 participants completed intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Karate Class Participants
Number analyzed (Participants) | 15
score on a scale | 19.3 (19.6)

4. Secondary Outcome: Attendance at Twice Weekly Classes
Description: Attendance at twice weekly classes, measured by karate instructors
Time Frame: Ten weeks
Measure: Mean (Standard Deviation); unit: percentage of classes attended
Arm/Group | Karate Class Participants
Number analyzed (Participants) | 15
percentage of classes attended | 86.7 (9.9)

5. Secondary Outcome: "Would You Recommend Karate Classes to Another Individual With Parkinson's Disease?"
Description: Number of individuals answering "Yes"
Time Frame: Ten weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Karate Class Participants
Number analyzed (Participants) | 15
Participants | 15

6. Other Pre Specified Outcome: Change in Balance Abilities as Measured by the Functional Reach Test (FRT)
Description: The Functional Reach Test (FRT) is a brief, valid, reliable, and practical assessment of balance. This test involves a yardstick being mounted on a wall at shoulder height. The subject is asked to stand next to the yardstick, extend the arm closest to the wall at 90 degrees of shoulder flexion, and the distance is recorded. The subject is then asked to reach as far as he or she can forward without taking a step, and the distance is recorded again. The difference between start and end position is the reach distance. Greater reach distances indicate better balance. Scores at the pre- and post-intervention focus groups will be compared.
Time Frame: 10 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Balance Abilities as Measured by the Tinetti Mobility Test (TMT)
Description: The Tinetti Mobility Test (TMT) consists of 2 subscales: balance tests (9 items, scored from 0-16) and gait tests (7 items, scored from 0-12), where higher scores reflect better performance. Scores at the pre- and post-intervention focus groups will be compared
Time Frame: 10 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Anxiety as Measured by the Hospital Anxiety and Depression Scale (HADS)
Description: The Hospital Anxiety and Depression Scale (HADS) is a brief, 14-item highly validated scale for measuring anxiety (7 items) and depression (7 items), where scores of >8 for either anxiety or depression indicate probable symptoms. Scores at the pre- and post-intervention focus groups will be compared.
Time Frame: 10 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Cognitive Abilities as Measured by the Symbol Digit Modalities Test (SDMT)
Description: In the Symbol Digit Modalities Test (SDMT), the subject uses a reference key to pair specific numbers with given abstract geometric figures in 90 seconds. Scores are the correct number of pairs made in 90 seconds, with greater scores indicating greater cognitive abilities. Scores at the pre-and post-intervention focus groups will be compared.
Time Frame: 10 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Short-term Memory Abilities as Measured by the Digit Span Test (DST)
Description: The Digit Span Test (DST) tests the number of digits a subject can recall in the correct order after hearing them. The experimenter says numbers slowly at one second intervals. Subjects are asked to repeat the numbers in the order they were given. A subject's digit span is the number of items they are able to report back in order correctly. Scores at the pre-and post-intervention focus groups will be compared.
Time Frame: 10 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Number of Participants Continuing to Attend Karate Classes
Description: During the six month follow-up phone call, subjects will be asked whether they have continued to participate in any structured karate or martial arts classes. If yes, frequency and location of these classes will be asked. If no, reasons for lack of participation will be asked. Larger numbers of "yes" responses would indicate program sustainability.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Karate Class Participants
Number analyzed (Participants) | 15
Participants | 8

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Karate Class Participants
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 1/19
Other Adverse Events (participants affected / at risk) | 1/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Karate Class Participants (N=19)
Appendicitis (Gastrointestinal disorders) | 1 (1) — Not deemed related to study
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Karate Class Participants (N=19)
Exacerbation of pre-existing sciatica (Nervous system disorders) | 1 (1) — One participant reported exacerbation of pre-existing sciatica that occurred during study time frame but outside of class

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/95/NCT03555695/Prot_SAP_000.pdf